CLINICAL TRIAL: NCT03971851
Title: Testing and Validation of a Novel Frailty Index in a Surgical Cohort
Brief Title: Validation of a Novel Frailty Index in Surgical Cohorts
Status: Completed | Type: Observational
Sponsor: University of Iceland (Other)
Responsible Party: Sponsor
Other Study IDs: FrailtyAndSurgery
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2019-11

CONDITIONS: Surgery--Complications; Anesthesia Morbidity; Perioperative Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low frailty: Frailty risk score less than 5
  Interventions: Other: Frailty risk groups
- Intermediate Frailty: Frailty risk score 5-15
  Interventions: Other: Frailty risk groups
- High frailty: Frailty risk score 15 and above
  Interventions: Other: Frailty risk groups

INTERVENTIONS:
Other: Frailty risk groups — Patients older than 65 will be separated into groups of varying frailty risk

SUMMARY:
This study will validate the utility of a novel frailty index that uses ICD diagnoses to call frailty severity in a surgical cohort of patients 65 and older

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years or older, undergoing any surgery at Landspitali University Hospital with an anesthesia team involved

Exclusion Criteria:

* No American Society of Anesthesiology classification provided

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals over 65 years of age undergoing surgery at a University Hospital Setting
Sampling Method: Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30-days
  Mortality within 30 days of surgery in each of the three frailty risk groups
Time to hospital readmission | Up to 180 days
  For patients surviving index hospitalization, the proportional hazard ratio of readmission between the three frailty group

SECONDARY OUTCOMES:
Long-term mortality | Up to 14 years
  Long-term mortality of the three different frailty risk groups, compared with proportional hazard modeling
Prolonged hospital length-of stay | 3 months
  Incidence of patients staying more than 10-days after surgery in the three frailty risk cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Martin I Sigurdsson, MD, PhD, Principal Investigator — University of Iceland

IPD SHARING:
Plan to Share IPD: No
Just summary data will be shared